CLINICAL TRIAL: NCT03699150
Title: Cardio-metabolic Risk Factors, Osteoporosis and Thrombus Embolic Assessment, Along Woman's Life: an Observational Retrospective Study
Brief Title: Cardio-metabolic Risk Factors, Osteoporosis and Thrombus Embolic Assessment, Along Woman's Life
Status: Completed | Type: Observational
Sponsor: Silvia Maffei (Other)
Responsible Party: Sponsor-Investigator, Silvia Maffei, Principal Investigator, Fondazione Toscana Gabriele Monasterio
Organization: Fondazione Toscana Gabriele Monasterio (Other)
Other Study IDs: 3605/2012
Record Dates: First submitted 2018-09-07; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Women's Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postmenopausal women: Outpatients referred to the Gynecologic Endocrinology, FTGM

SUMMARY:
Background: It is well known that health risks change during lifespan. The weight of a single risk factor increases with aging. The clinical significance of a single risk factor is clear but there is a lack on the effectof multiple risk factors linked together along different hormones condition of women's life in particular regarding to metabolic syndrome, osteoporosis, and thromboembolic risk.

Aim: 1) characterization and follow up of cardiometabolic risk in women of childbearing age; 2) characterization and follow up of cardiometabolic risk and osteoporosis in menopausal-transition women and in post-menopausal women;

DETAILED DESCRIPTION:
Background: It is well known that health risks change during lifespan. The weight of a single risk factor increases with aging. The clinical significance of a single risk factor is clear but there is a a lack on the effectof multiple risk factors linked together along different hormones condition of women's life in particular regarding to metabolic syndrome, osteoporosis, and thromboembolic risk. Moreover some pathological but reversible conditions during pregnancy may represent an incursion in metabolic syndrome and a sing of future cardiovascular disease.

Aim: 1) characterization and follow up of cardiometabolic risk in women of childbearing age; 2) characterization and follow up of cardiometabolic risk and osteoporosis in menopausal-transition women and in post-menopausal women; in outpatients referring to FTGM Ambulatory of cardiovascular gynecology and osteoporosis in Pisa.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients referred to the Gynecologic Endocrinology and Osteoporosis Unit of Fondazione CNR-Regione Toscana G. Monasterio, Pisa, Italy, who have authorized the use of their personal data

Exclusion Criteria:

* History of/or current neoplastic disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients referred to the Gynecologic Endocrinology and Osteoporosis Unit of Fondazione CNR-Regione Toscana G. Monasterio, Pisa, Italy.
Sampling Method: Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2012-06-22 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Effects of different contraceptive therapies on change of insulin sensitivity, lipidemic and inflammatory profile, coagulation and anthropometric parameters in fertile age women | Each patient is evaluated at t=0 (baseline) and after 3 months (t=1). To verify the permanence of change during also the follow up the same measures are repeated at 12 (T=2) months and then once a year (t=3, t=4) (when necessary)
  For each patient are collected data about:
  Oral glucose test tolerance (OGTT) with measures of glycemia (mg/dL) and insulinaemia (uU/mL) performed 7 times in 3 hours to obtain measure of insulin sensitivity (Matzuda-Index, OGIS Oral Glucose Insulin Sensitivity Index: (mL/min*m2)

SECONDARY OUTCOMES:
Effects of HRT and metabolic treatments on change of insulin sensitivity, lipidemic and inflammatory profile, coagulation, anthropometric parameters in menopausal transition and postmenopausal women. | Each patient is evaluated at t=0 (baseline) and after 3 months (t=1). To verify the permanence of change during also the follow up the same measures are repeated at 12 (T=2) months and then once a year (t=3, t=4) (when necessary)
  improvement of climacteric symptoms (Green Scale)
Effects of "bone therapies" on change of bone mineral density (BMD) in menopausal transition and post-menopausal women | Each patient is evaluated at t=0 (baseline) and after 3 months (t=1). To verify the permanence of change during also the follow up the same measures are repeated at 12 (T=2) months and then once a year (t=3, t=4) (when necessary)
  For each patient were collected:
  Bone DEXA: lumbar spine, total femoral (TF) and femoral neck (FN): BMD (g/cm2 ) of L1-L4, FN and TF BMD (g/cm2)
Effects of "bone therapies" on change of T-score in menopausal transition and post-menopausal women | Each patient is evaluated at t=0 (baseline) and after 3 months (t=1). To verify the permanence of change during also the follow up the same measures are repeated at 12 (T=2) months and then once a year (t=3, t=4) (when necessary)
  For each patient were collected:
  Bone DEXA: lumbar spine, total femoral (TF) and femoral neck (FN): T-Score L1-L4, T-Score FN, T-Score TF
Effects of "bone therapies" on change of Blood-markers of bone metabolism in menopausal transition and post-menopausal women | Each patient is evaluated at t=0 (baseline) and after 3 months (t=1). To verify the permanence of change during also the follow up the same measures are repeated at 12 (T=2) months and then once a year (t=3, t=4) (when necessary)
  For each patient were collected:
  Blood-markers of bone metabolism: Total Calcium(mmol/L), Ionized Calcium(mmol/L), alkaline bone phosphatase(ng/mL), Osteocalcin(ng/mL), Procollagen typeI, CTx(ng/mL), NTx(ng/mL), PTH(pg/mL), Vit D 25-OH(ng/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Maffei, MD, Principal Investigator — Fondazione Toscana Gabriele Monasterio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maffei S, Franchini M, Fortunato L, Guiducci L. Long-term effects of a combination of isoflavones, agnus castus and magnolia extracts on climacteric symptoms and cardiometabolic risk profile in postmenopausal women. Gynecol Endocrinol. 2022 Apr;38(4):339-344. doi: 10.1080/09513590.2022.2047171. Epub 2022 Mar 8. PMID 35257639
- [Derived] Guiducci L, Vassalle C, Parchi P, Maffei S. Monthly Intramuscular Neridronate for the Treatment of Postmenopausal Osteoporosis: Results of a 6-Year Prospective Italian Study. Int J Endocrinol. 2019 Feb 6;2019:9802827. doi: 10.1155/2019/9802827. eCollection 2019. PMID 30881452